CLINICAL TRIAL: NCT00310921
Title: A Randomized Study of Cervical Priming With Misoprostol Prior to Elective First Trimester Pregnancy Termination: Effects on Pain, Ease of Procedure and Complications
Brief Title: A Randomized Study of Cervical Priming With Misoprostol Prior to Elective First Trimester Pregnancy Termination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CN-00SFeig-04-B
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2005-11

CONDITIONS: Abortion, Therapeutic
MeSH Terms: interventions — Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
The purpose of this study is to determine whether misoprostol administered prior to elective first trimester pregnancy has an effect on pain and ease of procedure and complications.

DETAILED DESCRIPTION:
Previous studies suggest that cervical priming with misoprostol may facilitate vacuum aspiration for first trimester termination by inducing cervical dilation. This medication is used routinely at some abortion clinics, not at all at others and is used sporadically at most Kaiser facilities. The present study is designed to investigate whether the use of misoprostol noticeably improves the clinical experience. We will determine whether use of misoprostol compared with placebo during first trimester abortion 1) positively impacts ratings of pain experienced by the patient, 2) positively impacts physicians' ratings regarding difficulty of the procedure, and 3) reduces complications.

Misoprostol is effective for cervical priming prior to vacuum aspiration for first trimester pregnancy termination.2 Previous studies examined dose3,4, route of administration (oral5 or vaginal6,7) and time interval to allow maximum dilation while limiting side effects and bleeding prior to procedure.8,9,10 There is evidence supporting a specific dose, route and time interval.10 Previous studies also examined amount of bleeding, length of procedure, force used to dilate the cervix, and cervical dilation in mm.10 However, it is unknown whether these statistically significant changes translate into clinically relevant changes. For example, Ngai et al.10 report that the blood loss is significantly decreased. However, the mean blood loss differed at most by 68 ml. It is widely accepted that during surgical procedures a difference of 68 ml of blood will not change the patient's hematocrit or postoperative clinical course. In the same study preoperative baseline cervical dilation was only 1.7 mm different, also found to be statistically significant but there is no evidence that this difference changes the clinical experience for either the physician or the patient. All previous studies reviewed were also performed with the patient under general anesthesia so the patient's perception of pain was not examined. Because the majority of first trimester terminations in the U.S. are done with the patient awake, it is important to consider pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion criteria: after completion of a full history and physical exam each subject must be judged physically and mentally stable by the enrolling practitioner; subjects must be between 7 and 11 weeks pregnant and desiring termination. Gestation dating must be based on a reliable menstrual history consistent with a bimanual exam or ultrasound. All subjects must give informed consent after the study has been explained.

Exclusion Criteria:

* Subject must not have a physical or mental health condition which could be adversely affected by the study drug, including a history of allergy to prostaglandins or, specifically, to misoprostol.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2001-05; Study Completion 2006-05

PRIMARY OUTCOMES:
The first assessment will be a Visual Box Scale (VBS) for pain administered while the patient is undergoing the abortion procedure.

SECONDARY OUTCOMES:
After the procedure the physician will estimate the patient's pain using a VBS. The physician will also estimate the ease of the procedure using a different VBS.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Feigenbaum, M.D., Principal Investigator — Kaiser Permanente Medical Group, Inc.
Locations (1):
- Kaiser Permanente, Department of OB/GYN, San Francisco, California, United States